CLINICAL TRIAL: NCT01972763
Title: Ranibizumab for Recalcitrant Wet Age-related Macular Degeneration in Eyes Previously Switched From Bevacizumab and/or Ranibizumab to Aflibercept.
Acronym: RESCUE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northern California Retina Vitreous Associates (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28904
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Recalcitrant Wet Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

ARMS (2):
- Ranibizumab 1 mg (Active Comparator): Subjects will receive Ranibizumab 0.5 mg for 3 doses and then be separated into 2 arms based on initial response. In this Arm (Arm 1), patients will receive 1 mg of Ranibizumab monthly for the remainder of the study, if persistent or worse subretinal fluid with or without intraretinal cysts on SD-OCT is present.
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg (Active Comparator): Subjects will receive Ranibizumab 0.5 mg for 3 doses and then be separated into 2 arms based on initial response. In this Arm (Arm 2), patients will receive 0.5 mg of Ranibizumab monthly for the remainder of the study, if complete resolution of subretinal fluid on SD-OCT is present.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab is formulated as a sterile solution and will be used in the case of an intervention.

SUMMARY:
The purpose of the study is to determine the effectiveness of Ranibizumab 0.5 mg or 1.0 mg in subjects who were previously treated with Bevacizumab and subsequently switched to Aflibercept. These subjects have demonstrated a sub-optimal therapeutic response to the previous therapies; therefore, the study aims to see if Ranibizumab may have a greater treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age greater than or equal to 50 years
* Best-corrected ETDRS VA between 20/25 to 20/320
* Total area of subretinal hemorrhage and/or fibrosis comprising less than 50% of lesion
* Any neovascular lesion type of ARMD having previously received at least 3 doses 1.25 mg of bevacizumab and/or ranibizumab (minimum 3 monthly injections) followed by 3 monthly doses of aflibercept 2.0 mg (with last injection being within 8 weeks) with evidence of recalcitrant ARMD, defined by at least one of the following: persistent subretinal fluid with or without intraretinal cystic edema on SD-OCT and/or leakage on fluorescein angiography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation or pre-menopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* History of prior vitrectomy surgery
* Previous treatment with photodynamic therapy, radiation, or any other intravitreal drug delivery, such as dexamethasone or triamcinolone
* Subretinal hemorrhage involving the central fovea > 1 disc area, subfoveal atrophy
* CNVM secondary to causes other than ARMD
* Previous retinal pigment epithelial tear

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mean change in vision | 6 months

SECONDARY OUTCOMES:
Mean change in BCVA | 3 months, 9 months, and 12 months
Mean change in SD-OCT central foveal thickness | 3 months, 6 months, 9 months, and 12 months
Percentage of recalcitrant patients that respond by either OCT or VA to Ranibizumab after not having a complete response to previous therapy | 12 months
Percentage of patients that need to be escalated to 1 mg therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Wieland, MD, Principal Investigator — Northern California Retina Vitreous Associates
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States